CLINICAL TRIAL: NCT01605851
Title: GORE® Septal Occluder EU Clinical Evaluation: A Study to Evaluate Clinical Success and Performance in the Treatment of Transcatheter Closure of Patent Foramen Ovale (PFO)
Brief Title: GORE® Septal Occluder European Union Clinical Evaluation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: W.L.Gore & Associates (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GSO 11-05
Record Dates: First submitted 2012-05-18; First posted 2012-05-25 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Closure; Foramen Ovale
Keywords: PFO; closure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Closure, Foramen Ovale (Other): Patients undergoing device closure of PFO
  Interventions: Device: Closure, Foramen Ovale

INTERVENTIONS:
Device: Closure, Foramen Ovale

SUMMARY:
The primary objective of this study is to evaluate clinical success and performance of the GORE® Septal Occluder when used for percutaneous, transcatheter closure of Patent Foramen Ovale (PFO).

ELIGIBILITY:
Subjects with a PFO less than or equal to 17mm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2012-05; Primary Completion 2014-01 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
To evaluate clinical success and performance of the GORE® Septal Occluder when used for percutaneous, transcatheter closure of PFO | 6 months
  The primary endpoint for the study is composite Clinical Success evaluated at 6 months post-index procedure

SECONDARY OUTCOMES:
Additional Clinical Success evaluated during the procedure and 6 months post-procedure | 6 months
  Technical Success, Procedure Success, Closure Success

CONTACTS AND LOCATIONS:
Locations (9):
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet, Copenhagen
- Germany (4):
  - German Heart Center, Berlin
  - University Medical Center of Freiburg, Freiburg im Breisgau
  - Heidelberg University Hospital, Heidelberg
  - German Heart Center, Munich
- Hospital Group of San Donato, San Donato, Italy
- Karolinska University Hospital, Stockholm, Sweden
- Leeds Teaching Hospitals, Leeds, United Kingdom